CLINICAL TRIAL: NCT04502836
Title: Evaluation of the Correlation Between Psychological Intervention, Including Providing Knowledge and Tools for Problems Solving, and the Anxiety Level of Female Patients Arriving to ACTH LRH Test - Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: internal reasons
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RMC028220ctil
Record Dates: First submitted 2020-07-26; First posted 2020-08-06 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-03

CONDITIONS: Precocious Puberty
Keywords: ACTH LRH Test
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preliminary psychological intervention (Experimental): Participants in this group will receive a psychological intervention providing knowledge and tools for problems solving one hour prior to the ACTH LRH test.
  Interventions: Behavioral: Preliminary psychological intervention
- control group (No Intervention): Participants in this group will not receive any psychological intervention prior to the test.

INTERVENTIONS:
Behavioral: Preliminary psychological intervention — psychological intervention including providing knowledge and tools for problems solving according to the Choice - Agenda - Resilience - Emotional support (CARE) model . After intervention session patients and their parents will be asked to complete questionnaires
  Arms: preliminary psychological intervention

SUMMARY:
Over 20% of the population is reporting on "white coat syndrome", manifested as anxiety symptoms and elevated BP during interaction with medical staff. It is estimated that, throughout the life span of children, approximately 15-20% will suffer from some form of a trauma relating to an interaction with health provider. The proposed study aims is to evaluate the correlation between a single preliminary psychological intervention, including providing knowledge and tools for problems solving, and the anxiety level in female patients arriving to Adrenocorticotropic Hormone (ACTH) and Lutenising Releasing Hormone (LRH) test in comparison to the anxiety in patients arriving to the same test without psychological intervention. 20 female patients arriving to ACTH LRH test for puberty stage assessment (performed as part of routine medical care) will be recruited to the study and will be randomized to one of 2 groups. Participants in the intervention group (10 patients) will be required to arrive with their parents an hour prior to the test and will receive a preliminary psychological intervention. The control group will arrive to the ACTH LRH test on the scheduled time and will not receive psychological intervention

ELIGIBILITY:
Inclusion Criteria:

* Girls referred to ACTH LRH or LRH test
* Age 7-12 years old
* Ability to answer questionnaire independently (hebrew language only)

Exclusion Criteria:

* Mental disability
* Girls who were referred to the test in purpose of evaluation of the pituitary adrenal axis after prolong steroids therapy.
* Girls with chronic disease that required frequent hospitalization (over 4 times per year)

Ages: 7 Years to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Anxiety Questionnaire | Baseline (Visit 1), At the end of the ACTH LRH test, 2 hours

SECONDARY OUTCOMES:
Parents Treatment Satisfaction Questionnaire | Baseline (Visit 1), At the end of the ACTH LRH test, 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No